CLINICAL TRIAL: NCT06881472
Title: The Separate and Combined Glucagonotropic Effects of Glucose-dependent Insulinotropic Polypeptide and Alanine in Subjects With and Without Type 1 Diabetes
Acronym: GIPALANIN
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Asger Lund, MD (Other)
Responsible Party: Sponsor-Investigator, Asger Lund, MD, Associate professor, MD, Ph.D., University Hospital, Gentofte, Copenhagen
Organization: University Hospital, Gentofte, Copenhagen (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: H-21066812-113790
Record Dates: First submitted 2025-03-11; First posted 2025-03-18 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Type 1 Diabetes
Keywords: GIP; Amino acids; Alanine
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Incretins; Alanine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- GIP (Active Comparator)
  Interventions: Drug: Glucose-dependent Insulinotropic Polypeptide (GIP); Drug: Saline (NaCl 0,9 %) (placebo)
- Alanine (Active Comparator)
  Interventions: Drug: alanine; Drug: Saline (NaCl 0,9 %) (placebo)
- GIP + Alanine (Active Comparator)
  Interventions: Drug: Glucose-dependent Insulinotropic Polypeptide (GIP); Drug: alanine
- Placebo (Placebo Comparator)
  Interventions: Drug: Saline (NaCl 0,9 %) (placebo)

INTERVENTIONS:
Drug: Glucose-dependent Insulinotropic Polypeptide (GIP) — GIP
  Arms: GIP; GIP + Alanine
Drug: alanine — Alanine
  Arms: Alanine; GIP + Alanine
Drug: Saline (NaCl 0,9 %) (placebo) — Placebo
  Arms: Alanine; GIP; Placebo

SUMMARY:
The hormone glucose-dependent insulinotropic polypeptide (GIP) is naturally produced in the intestine during a meal and stimulates insulin secretion from the pancreas. Insulin ensures that nutrients from the meal are transported from the blood into the cells, allowing the body to use it as energy. If blood sugar levels drop too much, the body naturally releases another hormone: glucagon. Glucagon is responsible for the breakdown of nutrients inside the cells, thus causing blood sugar levels to rise again. This occurs, for example, when a person is fasting or in an energy deficit. Unfortunately, glucagon is not released in people with type 1 diabetes when blood sugar levels are low. However, it is known that GIP contributes to the secretion of glucagon during low blood sugar levels in both healthy individuals and those with type 1 diabetes.

Protein intake through the diet is broken down in the body into amino acids. It is known that the ingestion of protein and thus amino acids leads to an increase in glucagon in both healthy individuals and those with type 1 diabetes. This causes the amino acids to be converted into sugar, but also allows potentially harmful waste products from the breakdown to be converted into harmless components. The relationship between GIP and amino acids, as well as their joint effect on glucagon, is still unknown, but studies in mice have shown that if GIP and amino acids are given simultaneously, glucagon secretion will be even higher than if they were administered separately. The purpose of this study is to gain a better understanding of how the three (GIP, amino acids, and glucagon) are interconnected and affect each other and to see if the experiments conducted in mice yield the same results in healthy individuals and those with type 1 diabetes. Moreover, the secretion of glucagon, and thus the increase in blood sugar, might protect individuals with type 1 diabetes from experiencing low blood sugar. This knowledge could potentially be used for new treatment approaches in diabetes in the future.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian ethnicity
* Age between 18 and 70 years
* T1D (diagnosed according to the criteria of the World Health Organization) with HbA1c <69 mmol/mol (<8.5%)
* Body mass index between 20-27 kg/m2
* T1D duration of 2-20 years
* C-peptide negative (arginin-stimulated C-peptide ≤ 100 pmol/l)
* Treatment with a stable basal-bolus or insulin pump regimen for ≥3 months
* Informed and written consent

Exclusion Criteria:

* Anaemia (haemoglobin below normal range)
* Late microvascular complications except mild nonproliferative retinopathy
* Liver disease (alanine aminotransferase (ALAT) and/or aspartate aminotransferase (ASAT) >2 times normal values) or history of hepatobiliary disorder
* Treatment with any glucose-lowering drugs beside insulin
* Active or recent (within 5 years) malignant disease
* Active tobacco smoking / use
* Any condition considered incompatible with participation by the investigators

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only biological males, only cisgender men.
Enrollment: 10 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-01-16 (Estimated); Study Completion 2026-01-16 (Estimated)

PRIMARY OUTCOMES:
bsAUC of glucagon concentration | From 0-150 minutes
  Baseline Area under the curve of Glucagon concentration

SECONDARY OUTCOMES:
bsAUC Glucagon 30-90 | from 30-90 minutes
  Baseline corrected area under the curve of time spend in hyoglycaemia
bsAUC glucagon 90-150 min | from 90-150 minutes
  bs Glucagon in the recovery period

CONTACTS AND LOCATIONS:
Locations (1):
- Gentofte Hospital, Hellerup, Denmark